CLINICAL TRIAL: NCT00175539
Title: Group Psychoeducational Treatment for Women With Sexual Arousal Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05-0400
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Sexual Dysfunctions, Psychological
Keywords: sexual dysfunction; group treatment
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: psychoeducational intervention — three 1.5 hour long group psychoeducational sessions

SUMMARY:
The purpose of this study is to pilot test and determine the feasibility of a psychoeducational intervention (PED) we recently developed in a group format for women with acquired sexual arousal disorder (FSAD).

HYPOTHESES:

* 1 - Compared to baseline measures, the PED will result in significant improvement in self-report measures of: (a) subjective sexual arousal; (b) perception of genital arousal/genital sensitivity; (c) orgasmic experience; (d) sexual desire; (e) sexual distress; (f) relationship satisfaction; (g) depressive symptoms; and (h) quality of life.
* 2 - It is unknown what effect the PED will have on actual physiological sexual arousal.
* 3 - The group format will be a feasible and cost-effective method of delivering empirically supported treatment to women with sexual arousal difficulties and will contribute towards meeting the needs for sexual health care for women on the clinic wait-list at the BC Centre for Sexual Medicine.

DETAILED DESCRIPTION:
Sexual arousal difficulties are common among women, affecting approximately 22% of women between the ages of 18 and 59 (Laumann, Paik & Rosen, 1999). Although there are evidence-based psychological treatments available for women with orgasmic and pain disorders, there are currently no empirically-supported treatments for women with acquired Sexual Arousal Disorder (FSAD). Moreover, there have been numerous attempts to find evidence for a pharmacological agent effective at treating women's sexual arousal complaints; however, to date these studies have been inconclusive. Given the significant role that sexual health plays in quality of life, the fact that effective psychological treatments for women's sexual dysfunction are not widely available, and the fact that wait-lists to see health care professionals with expertise in the area of sexual dysfunction are often unwieldy, there is a need to establish brief, evidence-based approaches to treat women's acquired FSAD. Psychological therapy in a group format is a standard practice at the BC Centre for Sexual Medicine. However, in this study we would like to collect information from participants that would help us in determining the specific efficacy of the PED as well as identifying demographic or participant variables that might predict a positive response to the PED. Because we are using this information to determine the treatment's efficacy and because we will use this information as the basis for a publication, we deem this to be a research trial in which ethics review is necessary.

OBJECTIVES: We have recently developed and tested a new psychoeducational treatment (PED) for the treatment of FSAD due to early-stage gynecologic cancer treatment. Our data show this PED to significantly improve self-reported sexual desire, arousal, mood, relationship distress, and quality of life. We are currently testing the efficacy of this PED in a larger sample of cancer survivors with FSAD. The goal for this study is to test our PED in a group format for women who are currently seeking treatment at the BC Centre for Sexual Medicine for FSAD. By testing the efficacy of the PED administered in a group format, we hope to establish some preliminary data supporting the use of brief psychoeducational interventions for women. These pilot data will be used in a future larger-scale trial that involves randomization to group PED or a control condition in order to more definitively establish the PED efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 19 and 65 who are currently seeking treatment at the BC Centre for Sexual Medicine;
2. Women who are determined to meet criteria for acquired Female Sexual Arousal Disorder (FSAD);
3. Must be proficient in English and willing to take part in group sessions.

Exclusion Criteria:

Women who do not meet criteria for FSAD, as determined by the Co-Investigators, will not be informed about the study. In addition, women who might not be suitable for group therapy will be excluded.

-

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Upon completion of data analysis, establishment of the efficacy of Psychoeducational intervention (PED) in group format for the treatment women with Female Sexual Arousal Disorder will be determined. | following completion of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia
  - BC Centre for Sexual Medicine, Vancouver, British Columbia